CLINICAL TRIAL: NCT04011982
Title: PATAKESS Protocol : Clinical and Biological Analysis of Exocrine Pancreatic Tumors
Acronym: PATAKESS
Status: Recruiting | Type: Observational
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ET19-033 (PATAKESS)
Record Dates: First submitted 2019-06-20; First posted 2019-07-09 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Exocrine Pancreatic Cancer
Keywords: Pancreatic cancer; Immune infiltrate; Molecular alterations; Tumor stroma
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Exocrine pancreatic tumor samples (from initial diagnosis biopsy and/or from surgery specimen of primitive tumor and/or from metastases) and blood sample (collected during a routine check-up)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PATAKESS is a monocentric non interventional cohort study (prospective (alive patients) and retrospective (dead patients with biological material from surgery and/or biopsies already collected)).

PATAKESS consists of clinical and biological analyses of exocrine pancreatic tumors. Data are derived from tumor samples taken for routine health care purposes in patients managed at Centre Léon Bérard (Lyon-France) since January 2010. The main objective is to determine correlation between biological and clinical characterizations of patients suffering from exocrine pancreatic tumor.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma cancer is an aggressive cancer which represents 95% of pancreatic cancer. Pancreatic adenocarcinoma cancer is one of the deadliest cancers (5th cause of death per cancer) ; it has a very poor prognosis: 5-year survival (regardless of all stades at diagnosis). Pancreatic adenocarcinoma cancer is characterized by early metastasis. Therefore, development of efficient systemic therapeutics is one of the keys to improving prognosis. Newly developed immune check-point inhibitors seem to have limited efficacy in pancreatic adenocarcinoma except for MSI-H (Microsatellite instability-high) or dMMR (mismatch repair deficient)/MSI-H tumors.

However, recent data suggest that immune surveillance could control metastatic dissemination of pancreatic adenocarcinoma cancer. Several studies showed strong interactions between pancreatic tumor cells and tumor stroma in metastatic dissemination and in resistance to conventional therapeutics. Many data about pancreatic primitive tumors from murine animals models are available ; however few data on tumor stroma and its interactions with tumor cells of metastasis from adenocarcinoma pancreas are available. Few data on correlation between molecular alterations types (mutations, deletions, amplifications) in pancreatic adenocarcinoma cells and tumor stroma characteristics (primitive and metastatic stroma (cells composition, immune infiltration)) are also available.

In PATAKESS study, clinical and biological data are derived from tumor samples taken for routine health care purposes in patients managed at Centre Léon Bérard (Lyon-France) since January 2010.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient 18 age or older
* Patient operated on for exocrine pancreatic adenocarcinoma at Centre Léon Bérard since 01/01/2010.
* Histological diagnosis of exocrine pancreatic adenocarcinoma confirmed with surgery specimen.

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated on for exocrin pancreatic adenocarcinoma since January 1st, 2010.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Determination of the correlation between clinical characterizations and biological characterizations of patients suffering from exocrine pancreatic cancer | Up to 72 months
  Clinical characteristics of patients are consistent with tumor response at each treatment line and disease stage at diagnosis ; Biological characteristics will describe molecular alterations of the tumor by sequencing techniques like Next Generation Sequencing (NGS)

SECONDARY OUTCOMES:
Comparison of different tumor stroma : from surgery specimen of primitive tumor with preoperative chemotherapy, versus from surgery specimen of primitive tumor without preoperative chemotherapy, versus from biopsies done before chemotherapy | Up to 72 months
  Comparative characterization of the different stroma by immunological detection
Comparison of different tumor stroma : from surgery specimen of primitive tumor with preoperative chemotherapy, versus from surgery specimen of primitive tumor without preoperative chemotherapy, versus from biopsies done before chemotherapy | Up to 72 months
  Comparative characterization of the different stroma by NGS
Comparison of healthy tissu and tumor stroma from primitive tumor versus from metastases | Up to 72 months
  Comparative characterization of the different stroma by immunological detection
Comparison of healthy tissu and tumor stroma from primitive tumor versus from metastases | Up to 72 months
  Comparative characterization of the different stroma by NGS

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CASSIER, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France